CLINICAL TRIAL: NCT05642988
Title: Application of Wearable Technology in High-risk Surgical Patients in the Perioperative Period: a Feasibility Study
Brief Title: Application of Wearable Technology in High-risk Surgical Patients in the Perioperative Period
Status: Completed | Type: Observational
Sponsor: Mater Misericordiae University Hospital (Other)
Collaborators: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Pádraig Ó Scanaill, Consultant Anaesthetist, Mater Misericordiae University Hospital
Other Study IDs: 1/378/2207
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Adult ALL; Surgery; Anesthesia; Postoperative Complications
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult patients being discharged from hospital following intra-abdominal or pelvic surgery: Patient compliance with wearable biosensor monitoring after major intracavity surgery. The remote monitoring is made up of a wearable biosensor and a data-enabled relay device which will detect vital sign observations (ECG, heart rate, temperature and respiratory rate) and a health status assessment questionnaire.
  Interventions: Device: LifeSignals 1AX Biosensor

INTERVENTIONS:
Device: LifeSignals 1AX Biosensor — Biosensor worn by patients for 30-days after intra-abdominal or pelvic surgery on discharge from hospital

SUMMARY:
Unrecognised changes in patients' vital signs after surgery can result in preventable complications. Current standard practice includes routine monitoring of patient vital signs up until hospital discharge.

Upon discharge from hospital, all forms of routine vital sign monitoring ceases. The availability and use of wearable technology in healthcare is increasing rapidly. The role of wearable technology in the remote monitoring of patients at high-risk of post-operative complications and hospital readmission after discharge from hospital is unclear.

This pilot study is aimed to assess the feasibility of using wearable technology in patients recovering from major intracavity surgery after hospital discharge in the Irish healthcare setting.

DETAILED DESCRIPTION:
Patients undergoing major abdominal and pelvic surgery can have re-admission rates of over 20% in the first 90-days after surgery.

In Ireland the 30-day mortality following emergency abdominal surgery is 6.6%, and 90-day mortality 11.6% (1). Furthermore, 20% of post-operative deaths occur after hospital discharge in those over 80 years of age, of which over 95% occurs during the first six-weeks (2).

Despite this high risk, many patients are discharged home from hospital when medically fit and continuous monitoring discontinues. In hospital, patient monitoring is routine to identify patient deterioration at an early stage using the national early warning score (NEWS), which consists of the following clinical observations: heart rate, blood pressure, temperature, respiratory rate, oxygen saturation and level of consciousness. This monitoring is done routinely in the hospital ward at least every four hours. This monitoring stops when patients are discharged from hospital. Patients discharged are given general advice for recovery and, as part of current practice, are advised to contact their General Practitioner (GP) or emergency department if feeling unwell. Despite this, mortality in the post-discharge period accounts for nearly a quarter of all post-operative deaths.

Home monitoring of patients with chronic conditions has previously been shown to be of some utility. Recently, during the COVID-19 pandemic, remote home monitoring of patients diagnosed with COVID-19 who did not meet hospital admission criteria were managed by smartphone application and peripheral pulse oximetry.

To date, no previously published studies have adopted home monitoring for a patient group that is at a high risk of re-admission. In addition, simple questionnaires used to monitor postoperative recovery (such as the QoR-15) exist, that are reflective of a patient's current health status, but they have not been used to monitor patients after hospital discharge.

In this study, the investigators aim to test the feasibility and patient compliance of remote wearable biosensor technology monitoring after major intracavity surgery. The remote monitoring combines vital sign observations (ECG, heart rate, temperature and respiratory rate) and a health status assessment questionnaire.

The study protocol has been approved by the Mater Misericordiae University Hospital Institutional Review Board (IRB) (Reference: 1/378/2207). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Scheduled to undergo or recently undergone major intra-cavity abdominal surgery
* Able to give informed written consent to participate

Exclusion Criteria:

* Deemed unfit for surgery
* Unable or unwilling to comply with remote monitoring for any reason
* Unable or unwilling to fill in a questionnaire in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients recovering from major intra-cavity abdominal surgery being discharged from the Mater Misericordiae University Hospital in Dublin, Ireland.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Compliance with wearable technology | 30-days
  Assess compliance with remote monitoring in the first 30-days after hospital discharge following intra-abdominal or pelvic surgery. Compliance will be defined as wearing the biosensor for at least 20 hours per day.

SECONDARY OUTCOMES:
Unplanned hospital admission or GP visits | 30-days after hospital discharge
  Retrospectively review any unplanned hospital admissions or GP visits in the first 30-days after hospital discharge
Heart rate | 30-days after hospital discharge
  Retrospectively review variations in heart rate (beats per minute) in the first 30-days after hospital discharge
Temperature | 30-days after hospital discharge
  Retrospectively review variations in temperature (degrees celsius) in the first 30-days after hospital discharge
Respiratory Rate | 30-days after hospital discharge
  Retrospectively review variations in respiratory rate (breaths per minute) in the first 30-days after hospital discharge
Quality of recovery score (QoR15) | 30-days after hospital discharge
  This score can range from 0 - 150, with higher scores relating to a more favourable recovery from surgery. This will be performed at day 30 after hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Data for patients will strictly follow the agreed Data Protection Agreement (DPA) put in place by the Mater Misericordiae University Hospital